CLINICAL TRIAL: NCT05407272
Title: National Taipei University of Nursing and Health Sciences
Brief Title: Explore the Sharing Model Intervene to Improve the Knowledge, Attitudes, Service Intentions and Service Start-up Effects of the Eight Major Non-cancer Disease End-stage Caregivers on Well-being and Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wen-Shiou Pan (Other)
Responsible Party: Sponsor-Investigator, Wen-Shiou Pan, National Taipei University of Nursing and Health Sciences, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: WSPan
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Alzheimer Disease, Late Onset; Stroke; Heart Failure; Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis Pulmonary Exacerbation; Chronic Liver Disease and Cirrhosis; Kidney Failure, Acute; Kidney Failure, Chronic
Keywords: knowledge of palliative care service; attitude of palliative care service; intention of palliative care service; initiation of palliative care service; home care
MeSH Terms: conditions — Alzheimer Disease; Stroke; Heart Failure; Pulmonary Disease, Chronic Obstructive; Fibrosis; Acute Kidney Injury; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared mode intervention group (experimental group) (Experimental): Methods of collecting cases The subjects whose identity card numbers last in odd numbers are in the experimental group and even numbers are in the control group. They are randomly divided into two groups - the shared mode intervention group (experimental group) and the home care routine care group (control group). The experimental group was given a weekly sharing mode intervention for six weeks, 20-60 minutes per week; the control group was given the home health education manual in the third week.
  Interventions: Other: Health Education Manual
- home care routine care group (control group) (Active Comparator): Methods of collecting cases The subjects whose identity card numbers last in odd numbers are in the experimental group and even numbers are in the control group. They are randomly divided into two groups - the shared mode intervention group (experimental group) and the home care routine care group (control group). The experimental group was given a weekly sharing mode intervention for six weeks, 20-60 minutes per week; the control group was given the home health education manual in the third week.
  Interventions: Other: manual

INTERVENTIONS:
Other: Health Education Manual — A health education manual based on a shared model
  Arms: Shared mode intervention group (experimental group)
Other: manual — routine care
  Arms: home care routine care group (control group)

SUMMARY:
Since September 1st, 2009, Taiwan has begun to pay attention to the care of patients with organ failure, dementia and the elderly, and brought eight of non-cancer terminal patients into health insurance subsidies to implement the goal of universal palliative care and local aging. Taiwan has entered the aged society since March 2018, become the heavy burden of expenditure in Taiwan because of the health care needs and costs associated with the rapid aging of the population. With advanced medical technology, when facing inevitable death situation, should not use too much medical treatment on terminally ill patients. The waste of medical resources and bring both patients and family members so much pain. In Taiwan, people have misconception about tranquil palliative care. The low rate of home palliative care for non-terminal cancer patients. The purpose of this study is investigating the eight non-cancer terminal caregivers' knowledge, attitudes and service intentions of palliative care, and getting the result by research intervention.

In this study, a randomized experimental research design was applied by two-group pre-and post-test. The targets are the eight non-cancer terminal caregivers in a home care institution of a regional teaching hospital located in Yilan. Targets' ID end with odd numbers are in experimental group received shared mode intervention, and even numbers are in control group received home routine care. The experimental group was implementing measures of weekly shared mode intervention in 20 to 60 minutes for six weeks; the control group started to implement measures of home care medical instructions booklet in the third week. The content of the outcome measurement questionnaire includes: basic information of the eight non-cancer terminal caregivers, the palliative care knowledge scale, the palliative care attitude scale, and palliative care service initiation intention scale. Data were analyzed by statistical methods such as descriptive analysis, independent sample t-test, paired-samples t-test, Pearson correlation analysis and one-way ANOVA.

DETAILED DESCRIPTION:
The valid sample of this study consisted of 60 individuals, 31 females and 29 males, with a mean age of 56.3 years, and one attrition (death), with an attrition rate of 1.67%. The results showed that (1) there was a significant difference between the experimental group and the control group in the mean pre-test and post-test of hospice and palliative care knowledge (t=-4.973, p=0.00) and palliative attitude (t=-2.424, p=0.02). (2) There were significant differences in the pre-test and post-tests of hospice and palliative care knowledge (p=0.000), hospice and palliative care attitude (p=0.008), and hospice and palliative care intention (p=0.009) in the experimental group; there were significant differences in the pre-test and post-tests of hospice and palliative care knowledge in the control group (p=0.002). (3) There were significant differences in hospice knowledge, attitude, intention and hospice initiation between subjects in the experimental group with and without a signed DNR or ACP, indicating that those with a signed DNR or ACP had higher scores in hospice knowledge, attitude, intention and hospice initiation, which was a significant factor in the results of this study; there were significant differences in hospice knowledge and intention between the control group in terms of education level. This means that higher education level, higher score of hospice knowledge and intention. (4) After the shared model study intervention, 24 (72.7%) signed the DNR or ACP consent form and 16 (48.5%) initiated hospice services; after the home care routine care, 3 (11.1%) signed the DNR or ACP consent form and 0 (0%) initiated hospice services.

ELIGIBILITY:
Inclusion Criteria:

1. Caregivers of terminally ill patients with eight major non-cancer diseases diagnosed by a physician.
2. The caregiver must be at least 18 years old and literate.
3. The caregiver has a clear awareness and can communicate in Mandarin or Taiwanese

Exclusion Criteria:

1. Diagnosed by a physician as a terminally ill patient with eight major non-cancer diseases.
2. Clear awareness and able to communicate in Mandarin or Taiwanese.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
the knowledge, attitudes, service intentions and service start-up effects of the eight major non-cancer disease end-stage caregivers on well-being and palliative care | six weeks
  The content of the outcome measurement questionnaire includes: basic information of the eight non-cancer terminal caregivers, the palliative care knowledge scale, the palliative care attitude scale, and palliative care service initiation intention scale. Data were analyzed by statistical methods such as descriptive analysis, independent sample t-test, paired-samples t-test, Pearson correlation analysis and one-way ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: WEN-SHIOU PAN, Principal Investigator — National Taipei University of Nursing and Health
Locations (1):
- Wen-Shiou Pan, Yilan, Taiwan

IPD SHARING:
Plan to Share IPD: No